CLINICAL TRIAL: NCT03306199
Title: Turbo Power Laser Atherectomy Combined With Drug Coated Balloon Angioplasty for the Treatment of Femoropopliteal De Novo/ Restenotic and In-Stent Restenosis Lesions
Brief Title: TurboPower + DCB Treatment of Femoropopliteal De Novo/ Restenotic and In-Stent Restenosis Lesions
Status: Completed | Type: Observational
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-0906
Record Dates: First submitted 2017-10-05; First posted 2017-10-10 (Actual); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Laser Atherectomy — The Turbo-Power is a laser atherectomy catheter designed for treatment of de novo or restenotic lesions in native infrainguinal arteries and for the treatment of femoropopliteal artery in-stent restenosis (ISR) in bare nitinol stents with adjunctive percutaneous transluminal angioplasty (PTA).

SUMMARY:
A retrospective study to evaluate Turbo Power laser atherectomy + drug coated balloon (DCB) angioplasty for the treatment of femoropopliteal de novo/restenotic lesions and in-stent restenosis (ISR).

ELIGIBILITY:
Inclusion Criteria:

* All patients treated for femoropopliteal de novo/restenotic lesions or in-stent restenosis using Turbo Power laser atherectomy plus drug coated balloon angioplasty

Exclusion Criteria:

* Any incomplete data on procedural approach and treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are recruited from the investigator's general patient population, and they must meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Institute of the South, Houma, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Turbo Power + DCB: Study participants were included if they had been treated with Turbo Power atherectomy + DCB within the study timeframe.
Period: Overall Study
Arm/Group | Turbo Power + DCB
Started | 82
Completed | 67
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Turbo Power + DCB
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Target Lesion Revascularization (TLR)
Description: A Target Lesion Revascularization is defined as any percutaneous or surgical intervention to treat a restenosis or reocclusion in the target lesion
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Turbo Power + DCB
Number analyzed (Participants) | 67
Participants | 52

ADVERSE EVENTS:
Time Frame: 1 year
Description: TLR, Amputation and Death were collected out to 12 months post-procedure for this retrospective study. Other (Not including serious) adverse events were not captured in this study. Events were collected through review of patient charts within study period.
Arm/Group | Turbo Power + DCB
All-Cause Mortality (participants affected / at risk) | 2/67
Serious Adverse Events (participants affected / at risk) | 16/67
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turbo Power + DCB (N=67)
TLR (Vascular disorders) | 15 (15) — Target Lesion Revascularization
Death (Cardiac disorders) | 2 (2)
Amputation (Vascular disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT03306199/Prot_SAP_000.pdf